CLINICAL TRIAL: NCT02330731
Title: N-butyl-2-cyanoacrylate, Iso-amyl-2-cyanoacrylate and Hypertonic Glucose With 72% Chromated Glycerin in Gastric Varices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sara Abdelhakam, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 482
Record Dates: First submitted 2015-01-01; First posted 2015-01-05 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2015-01

CONDITIONS: Gastric Varices
MeSH Terms: conditions — Esophageal and Gastric Varices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- N-butyl-2-cyanoacrylate (Other): injection sclerotherapy for gastric varices
  Interventions: Procedure: injection sclerotherapy for gastric varices
- iso-amyl-2-cyanoacrylate (Other): injection sclerotherapy for gastric varices
  Interventions: Procedure: injection sclerotherapy for gastric varices
- 72% chromated glycerin (Other): injection sclerotherapy for gastric varices
  Interventions: Procedure: injection sclerotherapy for gastric varices

INTERVENTIONS:
Procedure: injection sclerotherapy for gastric varices — The intravariceal technique of injection

SUMMARY:
AIM: To compare between n-butyl-2-cyanoacrylate, iso-amyl-2-cyanoacrylate and mixture of 72% chromated glycerin with hypertonic glucose solution in management of gastric varices.

METHODS: Ninety patients with gastric varices presented to Endoscopy Unit of Ain Shams University Hospital were included. They were randomly allocated into three groups; each group included 30 patients treated with intravariceal sclerosant injections in biweekly sessions till complete obturation of gastric varices; Group I (n-butyl-2-cyanoacrylate; Histoacryl®), Group II (iso-amyl-2-cyanoacrylate; Amcrylate®) and Group III (mixture of 72% chromated glycerin; Scleremo® with glucose solution 25%). All the procedures were done electively without active bleeding. Recruited patients were followed up for 3 months.

DETAILED DESCRIPTION:
• Study Design & Sampling: This prospective randomized study is conducted on ninety patients with gastric varices presented to Endoscopy Unit of Ain Shams University Hospital. Patients with non-variceal causes for upper GIT bleeding and those with severe co-morbidity are excluded.

Patients are randomly allocated into three groups; each group includes 30 patients who will be treated with sclerosant injections in biweekly sessions till complete obturation of gastric varices, with follow up for 3 months:

* Group I (Histoacryl® Group),
* Group II (Amcrylate® Group) and
* Group III (Scleremo® with Glucose 25% Group). The three groups are matching as regards age, gender, cause of liver cirrhosis (viral hepatitis B or C), Child score and endoscopic findings (including number, grade of EV and size of GV).
* Tools of the study:

All included patients will be subjected to:

1. Complete clinical evaluation.
2. Laboratory investigations: CBC, liver profile, viral markers (HBs Ag, HB core Ab, HCV Ab) by ELISA technique.
3. Child classification according to the modified Child Pugh's criteria [13].
4. Abdominal ultrasonography: liver and spleen size, portal vein diameter and ascites.
5. Upper gastrointestinal endoscopy: using Pentax video endoscope EG 3440. Esophageal varices are classified according to their size at the gastroesophageal junction into 4 grades according to Westaby et al. [14].

   Gastric varices are classified into: gastro-esophageal varices (GEV) and isolated gastric varices (IGV) according to Sarin et al. [15].
6. Therapeutic interventions:

The intravariceal technique of injection is done according to Soehendra et al. [16].

Histoacryl® is diluted as 0.5 ml histoacryl: 0.8 ml lipidol as a contrast agent to dilute the adhesive material to fill the whole varix and to prevent rapid hardening and obstruction of the needle. The mixture is injected slowly to minimize the risk of embolization followed by injection of 2 ml of distilled water. The first ml of water is injected to push the material into the varix and the second ml is injected during withdrawal of the needle to prevent its obstruction [8].

Amcrylate® is injected slowly followed by injection of 2 ml distilled water without mixing with any other substances [17].

Scleremo® is mixed with glucose 25% in a ratio of 1:1. The mixture is injected very slowly and with the waiting for moments inside the variceal lumen after injection to give enough time for the sclerosing material to be in contact with the vessel wall that helps haemostasis. There is no need for distilled water injection [11].

Informed consent was obtained from all included patients and the study protocol was approved from the ethical guidelines committee.

All the procedures are done electively without active bleeding. The primary end point of this study is the obturation of gastric varices. The secondary endpoint is the occurrence of bleeding whether from the puncture site during or immediately after injection or delayed (in-hospital or after discharge) and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastric varices presented to Endoscopy Unit of Ain Shams University Hospital

Exclusion Criteria:

* Patients with non-variceal causes for upper GIT bleeding and those with severe co-morbidity

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2012-01; Primary Completion 2012-06 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
obturation of gastric varices | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Reda Elwakil, MD, Principal Investigator — Professor